CLINICAL TRIAL: NCT06241911
Title: Safety and Efficacy of Transcutaneous Auricular Vagus Nerve Stimulation in Patients With Narcolepsy Type 1: A Double-blind, Randomized, Sham-controlled Trial
Brief Title: Transcutaneous Auricular Vagus Nerve Stimulation in Patients With Narcolepsy Type 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liu Yonghong (Other)
Responsible Party: Sponsor-Investigator, Liu Yonghong, chief of neurology, Xijing Hospital
Organization: Xijing Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KY20222053-C-1
Record Dates: First submitted 2024-01-16; First posted 2024-02-05 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Narcolepsy Type 1; Fmri
Keywords: transcutaneous auricular vagus nerve stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tVNS (Active Comparator): transcutaneous vagus nerve stimulation on the left auricle with 25-Hz frequency, with a 30-second on/off cycle.
  Interventions: Device: transcutaneous auricular vagus nerve stimulation
- Sham tVNS (Sham Comparator): transcutaneous vagus nerve stimulation on the left earlobe with 25-Hz frequency, with the same stimulation parameters
  Interventions: Device: transcutaneous auricular vagus nerve stimulation

INTERVENTIONS:
Device: transcutaneous auricular vagus nerve stimulation — Transcutaneous auricular vagus nerve stimulation (tVNS) is a newly developed treatment for neuromodulation. It offers advantages such as being non-invasive, cost-effective, and not requiring battery changes, unlike invasive vagus nerve stimulation (iVNS). The auricular branch of the vagus nerve, which is the only afferent branch distributed on the surface of the human body, can be directly stimulated to produce effects similar to classic vagus nerve stimulation (VNS)

SUMMARY:
The study aimed to examine the efficacy and safety of tVNS as a complementary approach for NT1 by conducting a double-blind, randomized, sham-controlled trial. The specific objectives of the study were as follows: To evaluate the effects of complementary tVNS on the ability to maintain wakefulness, severity of narcolepsy, mood and quality of life in patients with NT1

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 12 years old with the ability to understand and complete the self-reported questionnaires
2. The patients met the international classification of sleep disorders third edition (ICSD-3) for NT126
3. Local residence for more than 3 months
4. Willingness to follow the trial plan as scheduled

Exclusion Criteria:

1. History of a clinically defined neurological or sleep disorders other than NT1
2. Any psychiatric disorder involving a history of psychosis
3. Any chronic condition affecting the ability to read or comprehend written instructions
4. Any substances abuse within the past 12 months
5. Pregnant or nursing
6. Metallic implants or devices contraindicating tVNS

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
maintenance of wakefulness test (MWT) | 12 weeks
  the changes in the maintenance of wakefulness test (MWT), mean sleep latency of the 4 MTW trials at baseline, week 4, week 8 and week 12, a clinical tool used to objectively measure the ability of patients with NT1 to maintain wakefulness and vigilance.

CONTACTS AND LOCATIONS:
Locations (1):
- Liu Yonghong, Xi'an, Shaanxi, China